CLINICAL TRIAL: NCT04316000
Title: Anxiety, Fear of Cancer and Quality of Life Degree Before and After Endoscopic Band Ligation Without Resection in Subepithelial Tumours of the Digestive Tract ≤15-mm Management: a Multicenter Prospective Study
Brief Title: Anxiety and Fear of Cancer Before and After Banding Without Resection in Small SET Management (QUALI-BANDING-SET)
Status: Suspended | Type: Observational
Why Stopped: Due to SARS-CoV2 (Covid-19) pandemia and its implications for outcomes bias.
Sponsor: Francesc Bas-Cutrina (Other)
Responsible Party: Sponsor-Investigator, Francesc Bas-Cutrina, Principal Investigator, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: QUALI-BANDING-SET
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Subepithelial Tumors
Keywords: Tumourophobia; Anxiety for Cancer; Quality of Life; Cancer Worry Scale (CWS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A - Removal of the Subepithelial Tumour: The subephitelial tumour is successfully removed by endoscopic band ligation without resection.
  Interventions: Other: Initial Anxiety and Fear of Cancer Test; Procedure: Endoscopic band ligation without resection of the subpetihelial tumour.; Other: 1-2 Months Anxiety and Fear of Cancer Test; Other: 1 Year Anxiety and Fear of Cancer Test
- B - Non Removal of the Subepithelial Tumour: The subephitelial tumour is not successfully removed due to various reasons (size >15-mm, not technical success,...).
  Interventions: Other: Initial Anxiety and Fear of Cancer Test; Other: 1-2 Months Anxiety and Fear of Cancer Test; Other: 1 Year Anxiety and Fear of Cancer Test
- C - Not Observed or Benign Subepithelial Tumour: The subephitelial tumour is not observed or is a benign entity, which does not require further interventions for these patients.
  Interventions: Other: Initial Anxiety and Fear of Cancer Test; Other: 1-2 Months Anxiety and Fear of Cancer Test

INTERVENTIONS:
Other: Initial Anxiety and Fear of Cancer Test — Answer to Hospital Anxiety and Depression Scale (HADS), Cancer Worry Scale (CWS) and European Five-Dimension Quality of Live test (EuroQol-5D) before the initial endoscopic procedure.
  Other Names: Initial Test
Procedure: Endoscopic band ligation without resection of the subpetihelial tumour. — Correct application of the elastic band in the subepithelial tumor, achieving its removal by self-amputation in the 4-6 weeks endoscopic ultrasonography (EUS) control.
  Other Names: Successful SET banding
  Groups: A - Removal of the Subepithelial Tumour
Other: 1-2 Months Anxiety and Fear of Cancer Test — Answer to Hospital Anxiety and Depression Scale (HADS), Cancer Worry Scale (CWS) and European Five-Dimension Quality of Live test (EuroQol-5D) after 1-2 months of the initial endoscopic procedure, knowing whether the tumor has either been removed or not, is a benign entity or has not been observed.
  Other Names: 1-2 Months Test
Other: 1 Year Anxiety and Fear of Cancer Test — Answer to Hospital Anxiety and Depression Scale (HADS), Cancer Worry Scale (CWS) and European Five-Dimension Quality of Live test (EuroQol-5D) after 1 year of the initial endoscopic procedure, knowing whether the tumor has either been removed or not.
  Other Names: 1 Year Test
  Groups: A - Removal of the Subepithelial Tumour; B - Non Removal of the Subepithelial Tumour

SUMMARY:
To analyze the hypothetical improvement in anxiety degree, quality of life and fear of cancer in patients diagnosed with a small gastrointestinal subeptithelial tumor when opting for the removal of the lesion.

DETAILED DESCRIPTION:
This "Quality of Life" study is directly related to the "BANDING-SET" study (NCT03247231), whose main aim is to analyze the effectiveness and safety of endoscopic band ligation without resection in the small gastrointestinal subepithelial tumours management.

Using three validated tests (Hospital Anxiety and Depression Scale [HADS], Cancer Worry Scale [CWS] and European Five-Dimension Quality of Live test [EuroQol-5D]) patients are evaluated before and after the endoscopic procedure.

Three main groups of patients are presented:

* GROUP A, in which the subephitelial tumour is successfully removed [hypothesis: anxiety and fear of cancer should decrease].
* GROUP B, in which the subephitelial tumour is not successfully removed due to various reasons (size >15-mm, not technical success,...) [hypothesis: anxiety and fear of cancer shuold be similar before-after].
* GROUP C, in which the subephitelial tumour is not observed or is a benign entity, which does not require further interventions for these patients [hypothesis: anxiety and fear of cancer should decrease].

ELIGIBILITY:
INCLUSION CRITERIA:

* Age between 18 and 80 years.
* Patient able to sign and understand the Informed Consent.
* Patient with a previously corroborated diagnosis of a subepithelial tumor (SET) by previous endoscopic ultrasonography (EUS), or possible diagnosis of SET by finding a subepithelial lesion (SEL) in a conventional endoscopy performed that will require a EUS study.
* Acceptance by the patient as a candidate of the BANDING-SET study (NCT03247231) of assessment of the effectiveness and safety of band ligation without resection of subepithelial tumors of the digestive tract ≤15-mm, with the prior signing of the Informed Consent of this study.
* Patient that understand the concept of the study and will complete all the time frame until the study end

EXCLUSION CRITERIA:

* No Informed Consent.
* No BANDING-SET study (NCT03247231) Informed Consent.
* Patients with functional diversity, unable to understand the nature and possible consequences of the study.
* Patients unable to maintain subsequent follow-up (lack of adherence).
* Patients with a life expectancy of less than 12 months.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with subepithelial lesions (SEL) in the gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Initial Anxiety degree | 1-2 months
  At 1-2 months, number of patients with a total anxiety score of 8 or more points in the Hospital Anxiety and Depression Scale (HADS), anxiety subescale.
  Hospital Anxiety and Depression Scale (HADS), anxiety subescale, legend:
  * 0-7 points: Normal.
  * 8-10 points: Borderline anxiety.
  * 11-21 points: Anxiety disorder.
Initial Fear of Cancer degree | 1-2 months
  At 1-2 months, number of patients with a total fear of cancer score of 11 or more points in the Cancer Worry Scale (CWS).
  Cancer Worry Scale (CWS) legend:
  * 6-10 points: Low.
  * 11-15 points: Moderate.
  * 16-20 points: High.
  * 21-24 points: Very high.

SECONDARY OUTCOMES:
Long-term Anxiety degree | 1 year
  At 1 year, number of patients with a total anxiety score of 8 or more points in the Hospital Anxiety and Depression Scale (HADS), anxiety subescale.
  Hospital Anxiety and Depression Scale (HADS), anxiety subescale, legend:
  * 0-7 points: Normal.
  * 8-10 points: Borderline anxiety.
  * 11-21 points: Anxiety disorder.
Long-term Fear of Cancer degree | 1 year
  At 1 year, number of patients with a total fear of cancer score of 11 or more points in the Cancer Worry Scale (CWS).
  Cancer Worry Scale (CWS) legend:
  * 6-10 points: Low.
  * 11-15 points: Moderate.
  * 16-20 points: High.
  * 21-24 points: Very high.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Bas-Cutrina, MD, Principal Investigator — Endoscopy Unit; Digestive Diseases Department; H. Universitari de Bellvitge.; Joan B Gornals, MD, PhD, Principal Investigator — Endoscopy Unit; Digestive Diseases Department; H. Universitari de Bellvitge.; Sebastià Videla, MD, PhD, Principal Investigator — Department of Clinical Pharmacology; H. Universitari de Bellvitge.
Locations (7):
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol (Can Ruti), Badalona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona, Catalonia
  - Hospital de Sant Pau i de la Santa Creu, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Catalonia
  - Hospital Universitari Joan XXIII de Tarragona, Tarragona, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390